CLINICAL TRIAL: NCT01479387
Title: Special Drug Use Investigation of Zevalin
Brief Title: Zevalin Post-marketing Surveillance for Adequateness of Image Interpretation Criteria in Japan
Acronym: ZEVALIN-SDUI
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Head Medical Development Japan, Bayer Yakuhin Co.LTD.
Other Study IDs: 15043
Record Dates: First submitted 2011-08-11; First posted 2011-11-24 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Non-Hodgkin's Lymphoma (NHL)
Keywords: Zevalin; CD20+; Non-Hodgkin's lymphoma; Mantle cell lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: [111]In-ibritumomab tiuxetan (Zevalin, BAY86-5128)

INTERVENTIONS:
Drug: [111]In-ibritumomab tiuxetan (Zevalin, BAY86-5128) — Patients who have received In-111 Zevalin.

SUMMARY:
This study is a regulatory post-marketing surveillance of Zevalin (ibritumomab tiuxetan) in Japan. In-111 Zevalin is, at first, injected to patient for gamma scan imaging to assess biodistribution of the Zevalin. When the imaging shows no altered distribution, Y-90 Zevalin is injected to the patient for the actual treatment. The objective of this study is to assess appropriateness and necessity of revision of the standardized criteria for image interpretation of In-111 Zevalin by comparing assessment by the investigator and the members of the committee for image interpretation of In-111 Zevalin. A total 40 patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received In-111 Zevalin to verify that expected biodistribution is present.

Exclusion Criteria:

* Patients who are contraindicated based on the product label.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population of this study is 40 patients who received In-111 Zevalin to access biodistribution of Zevalin.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2008-08; Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Assessment of abnormal distribution of In-111 Zevalin by the investigator [Two scales; Yes or No] | At 48-72 hours after In-111 Zevalin injection
Assessment of abnormal distribution of In-111 Zevalin by the central committee [Two scales; Yes or No] | At 48-72 hours after In-111 Zevalin injection

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Japan